CLINICAL TRIAL: NCT04174521
Title: Association Between Mother and Child Weight Gain: Statistical Methods With Validation
Status: Completed | Type: Observational
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other); University of Pennsylvania (Other)
Responsible Party: Principal Investigator, Bryan Shepherd, Professor of Biostatistics, Vanderbilt University Medical Center
Other Study IDs: 190557
Record Dates: First submitted 2019-11-20; First posted 2019-11-22 (Actual); Results first posted 2022-01-31 (Actual); Last update posted 2022-01-31 (Actual); Status verified 2022-01

CONDITIONS: Obesity, Childhood
MeSH Terms: conditions — Pediatric Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Mother-Child: Mothers who have delivered at VUMC and their children who are seen by Vanderbilt-affiliated physicians.

SUMMARY:
Using retrospective data from the Vanderbilt University Medical Center electronic health record, the investigators will study the association between mother's weight / weight change before and during pregnancy and the development of childhood obesity up until 5 years of age.

DETAILED DESCRIPTION:
The investigators are extracting de-identified retrospective data from the Vanderbilt University Medical Center electronic health record for mother-child pairs. From this data, the investigators will study the association between mother weight change during pregnancy and the risk of her child developing obesity during the first 5 years of life. Included mothers must have at least one weight measurement and at least one height measurement; they must have at least one child with weight/length measurements at birth and one additional same day height/weight measurement at or before 5 years of age.

ELIGIBILITY:
Inclusion Criteria:

* Mother-child pairs in the Vanderbilt University Medical Center (VUMC) electronic health record.
* The mothers must have at least one height measurement.
* The mothers must also have at least one weight measurement during pregnancy.
* The child must have birth length and weight measures and at least one same day height/weight measurement during their first 5 years of life.

Min Age: 0 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Mothers who have delivered at VUMC and their children who are seen by Vanderbilt-affiliated physicians.
Sampling Method: Non-Probability Sample
Enrollment: 20670 (Actual)
Dates: Start 2019-06-26 (Actual); Primary Completion 2021-08-01 (Actual); Study Completion 2021-08-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bryan Shepherd, PhD, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Mother-Child
Started | 20670 (A unit is defined as a mother-child pair; each unit was comprised of two participants: the mother and the child.)
Completed | 20670 (This was a retrospective observational study so there really was no drop-out.)
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Mother-child pairs meeting inclusion criteria, mothers and children are reported individually.
Arm/Group | Mother-Child
Number analyzed (Participants) | 20670
Age, Continuous [Median (Inter-Quartile Range); unit: years]
  Maternal Age at delivery | 28 [23.5 to 32.3]
  Child Age at delivery | 0 [0 to 0]
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Sex is reported separately for children and mothers.
  Participants
    Maternal sex: number analyzed (Participants) | 10335
    Maternal sex: Female | 10335
    Maternal sex: Male | 0
    Child sex: number analyzed (Participants) | 10335
    Child sex: Female | 4887
    Child sex: Male | 5448
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3082
  Not Hispanic or Latino | 17168
  Unknown or Not Reported | 420
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 154
  Asian | 1420
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4778
  White | 12778
  More than one race | 82
  Unknown or Not Reported | 1458
Region of Enrollment [Number; unit: participants]
  United States | 20670

OUTCOME MEASURES:

1. Primary Outcome: Obesity of the Child (in the Mother-child Pair) During the First 5 Years of the Child's Life
Description: Obesity of the child is defined as having a BMI-by-age classification greater than the 95th percentile based on the US CDC percentiles.
Time Frame: first 5 years of child's life
Measure: Count of Participants; unit: Participants
Groups:
- Mother-Child: Mothers-child pairs whose delivery occurred at VUMC and who are seen by Vanderbilt-affiliated physicians.
Arm/Group | Mother-Child
Number analyzed (Participants) | 10335
Participants | 1845

ADVERSE EVENTS:
Time Frame: Retrospective observational study; not applicable
Description: Retrospective observational study; not applicable. All-Cause Mortality, Serious, and Other (Not Including Serious) Adverse Events were not monitored/assessed.
Groups:
- Mother-Child: Mothers who have delivered at VUMC and their children who are seen by Vanderbilt-affiliated physicians. All-Cause Mortality, Serious, and Other (Not Including Serious) Adverse Events were not monitored/assessed.
Arm/Group | Mother-Child
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

LIMITATIONS AND CAVEATS:
This was a retrospective observational study, and subject to all of the usual challenges with that type of data (e.g., confounding and measurement error). The data provided here are extracted from the electronic health record and may be prone to errors. We performed an extensive chart review for a subset of 996 mother-child records and incorporated these validated data into analyses using statistical methods that account for measurement error.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-03-04): https://cdn.clinicaltrials.gov/large-docs/21/NCT04174521/Prot_SAP_000.pdf